CLINICAL TRIAL: NCT00005517
Title: Community Surveillance of Congestive Heart Failure
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5036; R01HL060959 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2005-11

CONDITIONS: Cardiovascular Diseases; Heart Failure, Congestive; Heart Diseases; Heart Failure
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure; Heart Diseases

SUMMARY:
To conduct a surveillance study of congestive heart failure (CHF).

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

Systematic surveillance was conducted of CHF among residents, 35-84 years old, of the Minneapolis-St.Paul metropolitan area (population 2.45 million, 1995 estimate) in two complementary domains: 1) hospitalization for CHF in two calendar years, five years apart (1995 and the year 2000); and 2) newly diagnosed CHF over a 9-year period (1993-2001) among members of a large Health Maintenance Organization (HMO). The magnitude and characteristics of hospitalized CHF were assessed in all 21 acute care hospitals of the metropolitan area. One-third of all discharges with ICD-9 CHF codes were sampled randomly (n about 5,000 per surveillance year), abstracted by trained nurses, and classified according to clinical criteria and the results of diagnostic tests. Newly diagnosed CHF was distinguished from recurrent episodes of decompensated CHF by thorough review of the hospital record. A complementary perspective on CHF, including the outpatient setting, was provided by a systematic study of members of HealthPartners, one of the largest HMOs in Minneapolis-St. Paul. Using the HealthPartners database, all newly diagnosed CHF cases between January 1, 1993 and December 31, 2001 (n about 1,900) were identified and the diagnosis validated. Beginning in January 1, 1999, newly diagnosed CHF cases were identified on an ongoing basis (n about 600), surveyed by mail, and followed for one-year from the original diagnosis. Surveillance of the HealthPartners population supplemented hospital surveillance and contributed data on incidence, prevalence, treatment, use of resources, and patient outcomes.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 35 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-08; Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Shahar — University of Minnesota

REFERENCES:
- [Background] Shahar E, Lee S, Kim J, Duval S, Barber C, Luepker RV. Hospitalized heart failure: rates and long-term mortality. J Card Fail. 2004 Oct;10(5):374-9. doi: 10.1016/j.cardfail.2004.02.003. PMID 15470646
- [Background] Goldberg RJ, Spencer FA, Farmer C, Meyer TE, Pezzella S. Incidence and hospital death rates associated with heart failure: a community-wide perspective. Am J Med. 2005 Jul;118(7):728-34. doi: 10.1016/j.amjmed.2005.04.013. PMID 15989906
- [Background] Goldberg RJ, Glatfelter K, Burbank-Schmidt E, Farmer C, Spencer FA, Meyer T. Trends in mortality attributed to heart failure in Worcester, Massachusetts, 1992 to 2001. Am J Cardiol. 2005 Jun 1;95(11):1324-8. doi: 10.1016/j.amjcard.2005.01.076. PMID 15904637